CLINICAL TRIAL: NCT06427590
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC47 Injection for Subcutaneous Use in Healthy and Obese Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASC47 in Healthy and Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ascletis Pharma (China) Co., Limited (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ASC47-101
Record Dates: First submitted 2024-05-10; First posted 2024-05-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-09

CONDITIONS: Chronic Weight Management
Keywords: ASC47

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SAD in healthy subjects-Cohort 1 (Experimental): SAD cohort 1, dose 1
  Interventions: Drug: ASC47; Drug: Matching placebo
- SAD in healthy subjects-Cohort 2 (Experimental): SAD Cohort 2, dose 2
  Interventions: Drug: ASC47; Drug: Matching placebo
- SAD in healthy subjects-Cohort 3 (Experimental): SAD Cohort 3, dose 3
  Interventions: Drug: ASC47; Drug: Matching placebo
- SAD in patients with obesity-Cohort 3A (Experimental): SAD Cohort 3A, dose 3
  Interventions: Drug: ASC47; Drug: Matching placebo

INTERVENTIONS:
Drug: ASC47 — single subcutaneous injection of ASC47
Drug: Matching placebo — single subcutaneous injection of Placebo

SUMMARY:
This will be a phase I, randomized, double-blind, placebo-controlled, single dose escalation study. This study will be conducted in three periods: the screening period, the treatment period, and the follow-up period.

This study aims to evaluate the pharmacokinetics and target engagement of ASC47 in healthy and obese subjects.

ELIGIBILITY:
Key inclusion Criteria:

* Subject have provided informed consent before initiation of any study-specific procedures
* Healthy male subjects or female subjects, between 18 and 55 years of age (inclusive).
* Females who are not pregnant or breastfeeding, or do not plan to become pregnant within 6 months and are willing to use effective contraceptive measures from the first dose of the investigational product until 3 months after the last dose are eligible.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and other screening procedures, eg.

Key exclusion Criteria:

* Have a clinically relevant acute or chronic medical condition or disease of the cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, or dermatologic systems as assessed by the investigator.
* Have any current or historical disease or disorder of the hematological system or significant liver disease or family history of bleeding/platelet disorders.
* Have a history of cancer (other than basal cell or squamous cell cancer of the skin which is fully excised), rheumatologic disease or blood dyscrasia.
* Have a history of febrile illness within 14 days prior to screening.
* Have a positive alcohol or drug screen at Screening or have a history of alcohol or drug abuse within the past 1 years.
* Have an autoimmune disease, is immunosuppressed or is in any way immunocompromised.
* Have used prescription drugs (other than hormone replacement therapy and medications for contraceptive purpose) within 14 days prior to the first dose of Investigational product.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 57 days
  Evaluate the incidence of Serious Adverse Events (SAEs) and Adverse Events (AEs) from after the first dose administration to 57 days.
ECG QT Interval | up to 57 days
  Evaluate the ECG QT Interval after single doses of ASC47.
Blood cell | up to 57 days
  Evaluate red blood cell count, white blood cell count and platelet count in liter (cells/L) after single doses of ASC47.
Hematology | up to 57 days
  Evaluate the levels of glucose, cholesterol, electrolytes after single doses of ASC47.

SECONDARY OUTCOMES:
AUC of ASC47 | up to 57 days
  Evaluate the Area under the plasma concentration versus time curve after single doses of ASC47.
Cmax of ASC47 | up to 57 days
  Evaluate the Peak Plasma Concentration after single doses of ASC47.
Cmin of ASC47 | up to 57 days
  Evaluate the Minimum Plasma Concentration after single doses of ASC47.
T1/2 of ASC47 | up to 57 days
  Evaluate the Terminal-Phase Half-Life after single doses of ASC47
CL/F of ASC47 | up to 57 days
  Evaluate the Apparent Systemic Clearance after single doses of ASC47.
Vd/F of ASC47 | up to 57 days
  Evaluate the Apparent Volume of Distribution after single doses of ASC47.
Lipid parameters | up to 57 days
  Evaluate the LDL-C, TG, TC, HDL-C after single doses of ASC47.

CONTACTS AND LOCATIONS:
Locations (1):
- Ascletis, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No